CLINICAL TRIAL: NCT01294579
Title: A Phase II Open-Label Study of Ofatumumab and Bendamustine Followed by Maintenance Ofatumumab for Indolent B-cell Non-Hodgkin's Lymphoma (B-NHL) Which Has Relapsed After Rituximab or a Rituximab Containing Therapy
Brief Title: Ofatumumab and Bendamustine Followed by Maintenance Ofatumumab for Rituximab Relapsed Indolent B-cell Non-Hodgkin's Lymphoma (B-NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 114612
Record Dates: First submitted 2011-02-03; First posted 2011-02-11 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's Lymphoma; Ofatumumab; Relapsed; Rituximab; Bendamustine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ofatumumab and bendamustine (Experimental): 1000 mg intravenous (IV) on day 1 of each cycle (cycles 1-6) for induction phase and 1000 mg IV every 2 months for 2 years.
  Bendamustine 90 mg/m2 was given on day 1 (after the ofatumumab infusion) and day 2 of each cycle (cycles 1-6)
  Interventions: Biological: Ofatumumab; Drug: Bendamustine

INTERVENTIONS:
Biological: Ofatumumab — 1000 mg intravenous (IV) on day 1 of each cycle (cycles 1-6) for induction phase
  1000 mg IV every 2 months for 2 years
Drug: Bendamustine — 90 mg/m2 on day 1 (after the ofatumumab infusion) and day 2 of each cycle (cycles 1-6)

SUMMARY:
The purpose of this phase II open label study was is to evaluate the safety and efficacy of ofatumumab and bendamustine followed by maintenance ofatumumab in subjects with indolent B-NHL who had relapsed after Rituximab treatment. A maximum of 53 subjects at least 18 years old with Small lymphocytic, lymphoplasmacytic, marginal zone lymphoma, or follicular lymphoma; Grades 1, 2 and 3a, would have been enrolled (34 in Stage 1 and 19 in Stage 2). Subjects should have had Rituximab-sensitive disease, defined as a Partial Remission (PR) or Complete Remission (CR) to the last rituximab-containing therapy lasting at least 6 months following completion of therapy or subjects should have relapsed or have had disease progression following response to prior rituximab-based therapy a Eastern Cooperative Oncology Group (ECOG) Performance status of 0 1 or 2. During the induction phase, ofatumumab 1000 mg IV on day 1 of each cycle (cycles 1-6) were followed by Bendamustine 90 mg/m2 IV on days 1, 2 of each cycle (cycles 1-6).During the maintenance phase, subjects with a PR or CR after the induction phase received ofatumumab 1000 mg IV every 2 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Small lymphocytic, lymphoplasmacytic, marginal zone lymphoma, and follicular lymphoma; Grades 1, 2 and 3a, defined according to World Health organization (WHO) guidelines. [Tefferi, 2008]
* Tumor was verified to be CD20+ (based on local evaluation), from a current or previous tissue biopsy. Tissue biopsy should be repeated if no report or specimen is available, CD20 staining was not previously performed, or there is clinical suspicion that the indolent lymphoma has transformed to aggressive lymphoma/higher malignancy grade.
* Rituximab-sensitive disease, defined as a Partial Remission (PR) or Complete Remission (CR) to the last rituximab-containing therapy lasting at least 6 months following completion of therapy. Last rituximab-containing therapy is defined as the last therapy regimen containing at least one full dose of rituximab.
* Relapse or disease progression following response to prior rituximab-based therapy, that requiried treatment by 2007 Revised Response Criteria for Malignant Lymphoma (RRCML) guidelines.
* CT imaging in screening (based on local evaluation) showing 2 or more clearly demarcated lesions with a largest diameter > 1.5 cm, or 1 clearly demarcated lesion with a largest diameter > 2.0 cm.
* ECOG Performance Status of 0, 1, or 2.
* Age ≥ 18 years.
* Life expectancy of at least 6 months in the opinion of the investigator.
* Women of childbearing potential must have had a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception during the study and for one year following the last dose of study drug.
* Men with a female partner of childbearing potential must have had either had a prior vasectomy or agree to use effective contraception from 2 weeks prior to administration of the first dose of study treatment until one year after the last dose of study treatment.
* Must not have been on any prohibited medications.
* Subjects who had received prior bendamustine were eligible if they had achieved a response (CR/PR) which lasted > 6 months after the end of bendamustine containing treatment.

Exclusion Criteria:

* Lactating women
* CLL, Grade 3b follicular lymphoma or evidence that the indolent lymphoma had transformed to aggressive lymphoma. Subjects suspicious for transformation should have undergone a biopsy to exclude the possibility of transformation. Subjects with a previous diagnosis of small lymphocytic leukemia (SLL) and a screening monoclonal B-lymphocyte count of ≥ 5000/µl are defined by 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria to have CLL; such patients were NOT eligible for this study.
* Rituximab-refractory disease, defined as failure to have responded to or progression within 6 months of completing rituximab or rituximab-containing combination therapy.
* Previous treatment with ofatumumab.
* Previous radioimmunotherapy (RIT) within 6 months of study entry. Subjects who have received RIT must have attained a PR or CR lasting at least 6 months, and must have recovered from any hematologic or other toxicity.
* Previous allogeneic stem cell transplantation at any time OR autologous stem cell transplantation within 6 months of study entry.
* Prior use of monoclonal antibody (other than anti CD20) within 3 months prior to randomization. Chemotherapy or other systemic lymphoma therapy within 4 weeks of study entry.
* Received treatment with an investigational agent within 4 weeks of study entry, or was actively participating in another interventional clinical study.
* Known Central Nervous System (CNS) involvement by lymphoma.
* Current or previous other malignancy within 2 years of study entry. Exception: Subjects who have been disease-free for 2 years or more, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Chronic or currently active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment including, but not limited to: chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, active Hepatitis C, and known HIV disease. All Human Immunodeficient virus (HIV)-positive subjects are excluded from this study, regardless of whether they have an Acquired Immunodeficiency Syndrome (AIDS) defining disease and/or are on antiviral therapy.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months of study entry, uncontrolled congestive heart failure, and uncontrolled arrhythmia. Subjects with congestive heart disease or arrhythmia such as atrial fibrillation whose cardiac disease is well controlled on a stable medical regimen are eligible.
* Other significant concurrent, uncontrolled medical conditions including, but not limited to, renal, hepatic, autoimmune, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which, in the Investigator's opinion, will impact study participation.
* Positive serology for Hepatitis B (HB) defined as a positive test for Hepatitis B surface antigen (HBsAg). In addition, if negative for HBsAg but (Hepatitis B core antibody (HBcAb) positive (regardless of Hepatitis B surface antibody [HBsAb] status), a HB DNA test had to have been performed and if positive the subject will be excluded. If HBV DNA is negative, subject may be included but must have undergone HBV DNA monitoring. Prophylactic antiviral therapy may have been initiated at the discretion of the investigator.
* Current active liver or biliary disease. Exception: Subjects with Gilbert's syndrome or asymptomatic gallstones, liver metastases related to indolent NHL or otherwise stable chronic liver disease per investigator assessment, are eligible.
* Screening laboratory values:

Neutrophils < 1.5 x 109/L (unless due to NHL involvement of the bone marrow). Platelets < 100 x 109/L (unless due to NHL involvement of the bone marrow). Serum creatinine ≥2.0 mg/dL; subjects with serum creatinine ≥2.0 mg/dL were are eligible if the creatinine clearance (Cockcroft Gault equation [Cockcroft, 1976]) is ≥40 mL/min.

Total bilirubin > 1.5 times ULN [upper normal limit] (unless due to liver involvement by NHL or Gilbert's disease).

Transaminases > 3 times ULN (unless due to NHL involvement).

* Known or suspected inability to fully comply with study protocol.
* Known or suspected hypersensitivity to ofatumumab, bendamustine or mannitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-05-17 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (22):
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Burbank, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Oxnard, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Orange Park, Florida
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Kettering, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, Vancouver, Washington
  - Novartis Investigative Site, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lyons RM, Shtivelband M, Kingsley E, Moezi M, Richards D, Sharman J, Feng X, Cannan M, Fellague-Chebra R, Boyd TE. Efficacy and safety of ofatumumab and bendamustine followed by ofatumumab maintenance in patients with relapsed indolent non-Hodgkin lymphoma after prior rituximab. Leuk Lymphoma. 2021 Jun;62(6):1353-1360. doi: 10.1080/10428194.2020.1869957. Epub 2021 Jan 15. PMID 33448893

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects completed represents subjects who completed treatment.
Period: Overall Study
Arm/Group | Ofatumumab and Bendamustine
Started | 49
Completed | 14
Not Completed | 35
Not completed — Disease progression | 12
Not completed — Adverse Event | 11
Not completed — Study closed/terminated | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African heritage | 3
  White | 45
  Mixed race | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate of Induction Therapy After Cycle 6 (28 Days) (FAS)
Description: Complete response (CR) included all of the following: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. All target nodes had to have regressed to ≤ 1.5cm in the longest diameter. Non-measureable nodes 1.1 to 1.5cm in the longest diameter and >1cm in the short axis at baseline had to regress to ≤ 1cm in the short axis by visual estimation; enlarged spleen or liver (with nodules) must have returned to normal size and nodules disappeared and if bone marrow was involved, infiltrate had to have cleared on repeat biopsy sample. CR was not valid without imaging data. The corresponding 2-sided 95% exact confidence interval (CI) of the response rate was estimated by the Clopper-Pearson method.
Time Frame: Baseline up to 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
percentage of participants | 24.5 [13.3 to 38.9]

2. Secondary Outcome: Overall Response Rate (ORR) During Induction Phase After Cycle 6 (FAS)
Description: The overall response = CR (defined in Primary Outcome) + Partial Response (PR) which required all of the following: > or = to 50% decrease from baseline in target nodules; > or = to 50% decrease in hepatic/splenic nodules and no increase in liver or spleen size; no unequivocal progression in non-target lestions; no new sites of disease.
Time Frame: Baseline up to 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
percentage of participants | 67.3 [52.5 to 80.1]

3. Secondary Outcome: Conversion Rate of Partial Response in Induction Phase to Complete Response With Maintenance Ofatumumab (FAS)
Description: Rate of conversion from PR in the Induction phase, to CR with maintenance ofatumumab in subjects who have a PR with induction therapy with ofatumumab and bendamustine
Time Frame: Partial response in induction phase up to 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 16
percentage of participants | 37.5 [15.2 to 64.6]

4. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) up to 30 Months (FAS)
Description: Progression free survival (PFS) is defined as the interval between first treatment and disease progression or death due to any cause. PFS criteria: A previously normal node (≤ 1.5 x ≤ 1.0cm), including nodes that were not previously visible, must increase to >2.0 x ≥ 1.5cm; ≥ 50% increase from nadir in the PPD of any target node. The long axis must increase by at least 5 mm and to >2.0cm.; ≥ 50% increase from nadir in the long axis of any target node. The long axis must increase by at least 5 mm and to >2.0 cm.; ≥ 50% increase from nadir in the SPD of target nodes and at least one node should have a long axis >1.5 cm.
Time Frame: Baseline up to approximately 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
percentage of participants
  PFS events | 42.9
  PFS events - Progression | 32.7
  PFS events - Death | 10.2
  censored - follow-up ended | 57.1

5. Secondary Outcome: Kaplan-Meier Estimates of Progression Free Survival up to 30 Months (FAS)
Description: Progression Free Survival (PFS) is defined as the interval between first treatment and disease progression or death due to any cause. PFS events: progression documented between scheduled visits, death before first PD assessment (or death at baseline or prior to any adequate assessments), death between adequate assessment visits. For the PFS analysis, the survival function was estimated using Kaplan-Meier estimates.
Time Frame: Baseline up to approximately 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
months | 29.7 [17.3 to NA] — Upper limit of CI was not estimable

6. Secondary Outcome: Pharmacokinetic Profile Which Includes Measuring Blood Levels of Ofatumumab and Bendamustine in Combination and Ofatumumab Alone During Maintenance Treatment and Measuring Blood Levels of Circulating B Cell
Description: Due to recruitment issues, this data analysis was not done per changes in planned analysis. This data was only presented as patient listings. The statistical analysis plan was modified to indicate that Pharmacokinetic/Pharmacodynamic exploratory analyses were not done.
Time Frame: up to 30 months
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 0

7. Secondary Outcome: All Deaths by Preferred Term (Safety Set) up to Approximately 30 Months
Description: Deaths were collected and were considered to be an on treatment death up to 60 days post treatment.
Time Frame: Baseline up to approximately 30 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 49
participants
  Disease progression | 3
  Pneumonia | 1
  Myelodysplastic syndrome -reported post study | 1
  Squamous cell carcinoma of lung | 1
  Chronic obstructive pulmonary disease | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 30 months
Description: Deaths are reported as a secondary outcome
Groups:
- Ofatumumab + Bendamustine: Ofatumumab + Bendamustine
Arm/Group | Ofatumumab + Bendamustine
All-Cause Mortality (participants affected / at risk) | 7/49
Serious Adverse Events (participants affected / at risk) | 18/49
Other Adverse Events (participants affected / at risk) | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Bendamustine (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 3
Anaphylactic reaction (Immune system disorders) | 1
Diverticulitis (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Bendamustine (N=49)
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 7
External ear pain (Ear and labyrinth disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 10
Chest discomfort (General disorders) | 3
Chills (General disorders) | 4
Fatigue (General disorders) | 30
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 3
Pyrexia (General disorders) | 8
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 12
Blood creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 7
Pollakiuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7
Night sweats (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Urticaria (Skin and subcutaneous tissue disorders) | 10
Flushing (Vascular disorders) | 5
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
The study was terminated early based on the evolution of the current therapeutic treatment landscape in Non Hodgkin Indolent Lymphomas and low enrollment rates for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.